CLINICAL TRIAL: NCT01194427
Title: A Multi-Institutional Phase II Study Evaluating Surrogate Biomarkers of Response to Short Term Oral Vorinostat and Tamoxifen in Women With Newly Diagnosed Breast Cancer
Brief Title: A Study of Vorinostat and Tamoxifen in Newly Diagnosed Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty meeting patient accrual goals
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: J09144; NA_00033768 (Other: Johns Hopkins)
Record Dates: First submitted 2010-03-25; First posted 2010-09-03 (Estimated); Results first posted 2013-05-17 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Stage I Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer; Invasive Breast Cancer
Keywords: Preoperative; Neoadjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — Vorinostat; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vorinostat and Tamoxifen (Experimental): Vorinostat and tamoxifen are taken for about 14 days prior to definitive surgery.
  Interventions: Drug: Vorinostat and Tamoxifen

INTERVENTIONS:
Drug: Vorinostat and Tamoxifen — vorinostat 400 mg PO once daily and tamoxifen 20mg PO once daily for 14 days
  Other Names: Zolinza

SUMMARY:
This research study is designed to look at the effects of the combination of vorinostat (Suberoylanilide Hydroxamic Acid or Zolinza) and tamoxifen on breast cancer tissue. The investigators will do this by comparing tissues from the original breast biopsy to tissues obtained after taking vorinostat and tamoxifen for 2 weeks.

DETAILED DESCRIPTION:
Key eligibility criteria include:

* Newly diagnosed invasive breast cancer awaiting surgery or neoadjuvant (preoperative) treatment
* No use of hormone contraceptives or replacement therapy within 30 days prior to the diagnostic breast cancer biopsy (unless willing to have an additional biopsy prior to starting the study)
* No prior or current use of any therapy to treat the current breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III invasive breast cancer
* Awaiting surgery or neoadjuvant treatment
* ECOG performance status 0, 1 or 2
* Adequate organ function
* Prior use of hormone contraception or replacement therapy must have been discontinued at least 30 days prior to diagnostic biopsy (unless participant is willing to undergo an additional biopsy for the study)

Exclusion Criteria:

* Prior or current treatment of any kind for the current breast cancer
* Current use of any other investigational drugs
* Uncontrolled or active infection, congestive heart failure, cardiac arrythmia, or psychiatric illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, M.D., Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be recruited through the breast cancer clinics at each of the participating centers (ie, Johns Hopkins).
Pre-assignment Details: Women 18 years or older with a histologically confirmed diagnosis of invasive mammary carcinoma on a core needle biopsy and with adequate organ function who are awaiting a definitive surgical procedure or initiation of neoadjuvant chemotherapy are eligible.
Period: Overall Study
Arm/Group | Vorinostat and Tamoxifen
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vorinostat and Tamoxifen
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Changes in Markers of Proliferation Prior to and After Study Drug Administration
Description: To determine the percentage change in proliferation index Ki-67 in both ER-positive and ER-negative tumors between baseline and post-treatment biopsy following 14 days of vorinostat 400 mg PO once daily and tamoxifen 20mg PO once daily in women with primary breast cancer awaiting definitive surgery.
Time Frame: Baseline and 14 days
Population: Two (2) participants were enrolled; however, due to difficulty in recruitment, we were not able to complete the study. There were not study-specific analyses completed or results to report.
Arm/Group | Vorinostat and Tamoxifen
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 14 days
Description: Adverse events were assessed at baseline, after 14 days of study drug administration, and after the surgical procedure per CTCAE V. 4.0.
Arm/Group | Vorinostat and Tamoxifen
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat and Tamoxifen (N=2)
Anorexia (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Unable to recruit participants to complete the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No